CLINICAL TRIAL: NCT05544760
Title: CatchU: A Quantitative Multisensory Falls-Assessment Randomized Clinical Trial
Brief Title: CatchU: A Quantitative Multisensory Falls-Assessment Study
Acronym: CatchU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Burke Rehabilitation Hospital (Other); Montefiore Medical Center (Other); Jet Worldwide Enterprises Incorporated (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-13418
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Fall Injury; Age Problem; Well Aging; Sensory Disorders
Keywords: falls; aging; multisensory integration
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial, first examines whether participants are good or bad multisensory integrators. If eligible and interested in participating, we will screen 300 participants level of multisensory integration. If participants are good integrators, no randomization will be necessary as these participants will not meet inclusion trial for the intervention trial. If participants are poor integrators, then they will be randomized into either the control (regular care) or intervention (CDC recommendations and falls counseling) arms. Note that be expect ~134 participants to be poor integrators. Those that are good integrators will not be included in the intervention trial but will be included in the larger observational study to test other study aims including 1) demonstrating acceptable concurrent validity of CatchU for identifying older adults' multisensory integration performance in older adults and 2) Examining predictive validity of CatchU in older adults.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Placement into the intervention vs. control group is random, but dependent upon multisensory integration performance. Meaning, older adults who are enrolled and screened with good integration abilities on the CatchU test (aka: VSI + (good) integrators), (VSI = visual-somatosensory integration) will not be placed in either the intervention or control group since better visual-somatosensory integration performance has been linked to better cognitive and motor outcomes. These participants will be included in examination of additional study aims not related to the intervention.
  VSI - (poor) integrators, will be randomly assigned into either the intervention or control group to test the beneficial effect of the CatchU intervention.
  Participants in the Control arm will be monitored every two months via telephone surveys to determine falls history, but will not receive the CatchU intervention.
- CatchU Intervention (Experimental): Placement into the intervention vs. control group is random, but dependent upon multisensory integration performance.
  VSI - (poor) integrators, will be randomly assigned into either the intervention or control group to test the beneficial effect of the CatchU intervention. Participants in the Intervention arm will be monitored every two months to determine falls history, but will also receive the CatchU intervention which consists of physicians relaying individualized recommendations from the CatchU physician report to the participant, as well as providing the participant with falls intervention referrals and falls counseling.
  Interventions: Other: CatchU Intervention

INTERVENTIONS:
Other: CatchU Intervention — The CatchU Intervention arm will receive individualized recommendations (adapted from the CDC STEADI program) as outlined on the CatchU physician report sent to the participants physicians. These recommendations in combination with falls intervention referrals and falls counseling tips will be monitored and statistical investigation of the impact of CatchU intervention in preventing future falls will be determined.
  Arms: CatchU Intervention

SUMMARY:
The ability to successfully integrate information across sensory systems is a vital aspect of functioning in the real world. To date, only a few studies have investigated the clinical translational value of multisensory integration processes. Previous work has linked the magnitude of visual-somatosensory integration (measured behaviorally using simple reaction time tasks) to important cognitive (attention) and motor (balance, gait, and falls) outcomes in healthy older adults. While multisensory integration effects have been measured across a wide array of populations using various sensory combinations and different neuroscience approaches, a gold standard for quantifying multisensory integration has been lacking. The investigator recently developed a step-by-step protocol for administering and calculating multisensory integration effects in an effort to facilitate innovative and novel translational research across diverse clinical populations and age-ranges. However, patients with severe medical conditions and/or mobility limitations often experience difficulty traveling to research facilities or joining time-demanding research protocols. Using the aforementioned protocol, the study team invented a mobile multisensory falls-assessment iPhone app called CatchU to facilitate physician discussion and counseling of falls in older adults during clinical visits (e.g., annual wellness visits with a subsequent telehealth call), in an attempt to alleviate disability, promote independence, and increase quality of life for older adults. The investigator team has provided a cross-sectional research proposal for a pilot study of 300 patients (over a 24-month period) in order to demonstrate acceptable-to-excellent predicative accuracy of CatchU for identifying older adults at-risk for falls.

ELIGIBILITY:
General inclusion criteria:

1. Adults aged 65 and older, residing in New York Metropolitan area who plan to be in area for next three or more years.
2. Able to speak English at a level sufficient to undergo our assessment battery.
3. Ambulatory. Participants are classified as 'non-ambulatory' if they are unable to leave the confines of their home and attend a clinic visit. These include participants who are bed-bound as a result of severe medical illness or those who require assistive medical devices (respiratory support or ventilators) that cannot be transported or those who cannot complete our mobility protocols. We will not exclude participants who use walking aids (canes, crutches) for ambulation. Participants who require walking aids to walk outside but are able to complete our mobility protocols without an assistive device or the assistance of another person will not be excluded.

General exclusion criteria (one or more criteria):

1. Presence of dementia as defined as a score of ≥ 2 on the Alzheimer's Disease 8 (AD8) or < 25 on The Montreal Cognitive Assessment (MoCA). These cut scores and procedures have been validated in our and other aging studies.
2. Serious chronic or acute illness such as cancer (late stage, metastatic, or on active treatment), chronic pulmonary disease on ventilator or continuous oxygen therapy or active liver disease. Individuals with recent cardiovascular or cerebrovascular event (Myocardial Infarction, Percutaneous Transluminal Coronary Angioplasty, Coronary Artery Bypass Graft, or stroke) will not be excluded if they meet above inclusion criteria. Many of these chronic conditions are very common in older adults. Hence, mere presence of these conditions will not be used to exclude participants if well controlled or of mild severity and if participants are able to complete training and mobility tasks.
3. Mobility limitations solely due to musculoskeletal limitation or pain (e.g., severe osteoarthritis) that prevent participants from completing mobility tests.
4. Any medical condition or chronic medication use (e.g., neuroleptics) in the judgment of the screening clinician that will compromise safety or affect cognitive functioning or terminal illness with life expectancy less than 12 months.
5. Progressive, degenerative neurologic disease (e.g., Parkinson's disease or ALS) diagnosed by study clinician or as per medical history.
6. Presence of clinical disorders that overtly alter attention like delirium.
7. Hospitalized in the past 6 months for severe illness or surgery that specifically affects mobility (e.g., hip or knee replacement) and that prevent participants from completing mobility tests or plans for surgery affecting mobility in the next 6 months.
8. Severe auditory, visual, or somatosensory self-reported impairments. Visual acuity will be screened using a Snellen chart by the psychological assistant. Presence of neuropathy will be assessed using the Michigan Neuropathy Screening Instrument.
9. Active psychoses or psychiatric symptoms (such as agitation) noted during the clinic visit that will prevent completion of study protocols. Past history of these symptoms or presence of psychiatric illness not used as exclusion criteria.
10. Living in nursing home.
11. Participation in another intervention trial. Participants can participate in other observational studies.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Falls | 24 months
  Information about falls (answers to questions regarding whether the participant has had a fall in the past 1 year or past 2 months after study enrollment) will be collected. If a fall is endorsed during the interview, further information regarding when and where the fall occurred and whether it led to a major injury or hospitalization will also be collected.
  The relationship of multisensory integration performance on CatchU with history of falls in the past year (baseline) and incident falls over a 24-month period post-baseline visit (collected bimonthly through telephone interviews) will be assessed using Cox proportional hazard models. Here we will look at fall presence (yes or no) and time to fall (or censor if no fall) relative to baseline enrollment date

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette R Mahoney, PhD, Study Chair — Albert Einstein College of Medicine; Mooyeon Oh-Park, MD, Principal Investigator — The Burke Rehabilitation Hospital
Locations (1):
- Burke Rehabilitation Hospital, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Investigator will determine whether participant data will be shared towards the conclusion of the study.

REFERENCES:
- See also: Catchu Website — http://catchu.net